CLINICAL TRIAL: NCT06391619
Title: Huntington's Disease Young Adult Study 2.0
Acronym: HD-YAS
Status: Active, not recruiting | Type: Observational
Sponsor: University College, London (Other)
Collaborators: University of Iowa (Other); University of Cambridge (Other); University of Glasgow (Other)
Responsible Party: Sponsor
Other Study IDs: 145646
Record Dates: First submitted 2024-01-26; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Huntington's disease gene carriers: Individuals with a positive test for the HD gene who were more than 20 years from expected symptom onset at baseline assessment.
  Interventions: Other: No intervention
- Controls: Healthy controls matched to the gene carrier group for age, sex and education
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Study is observational

SUMMARY:
The goal of this observational study is to learn about the first signs of disease in young adult carriers of the gene for Huntington's disease. The main questions to answer are:

* what are the earliest signs of the disease?
* can we identify the best time to intervene with treatment to prevent or delay onset of symptoms?
* can we identify the most reliable markers of disease for use in prevention trials?

Participants will undergo the following assessments:

* clinical examination
* cognitive and neuropsychiatric testing
* brain imaging
* biofluid sampling

Researchers will compare gene carriers with matched controls to see if any of these measures show evidence of early disease effects.

DETAILED DESCRIPTION:
We will undertake follow up assessments of the HD-YAS cohort comprising far-from-onset premanifest mutation carriers (preHD) (n=64) and controls, matched for age, sex and education (n=67). These assessments will occur approximately 4.5 and 6 years after their baseline assessment. They will include

* detailed clinical assessment
* cognitive testing using CANTAB and the EMOTICOM
* neuropsychiatric assessment
* neuroimaging including 3T volumetric MRI, NODDI, resting state fMRI and multiparametric mapping. A subset of 20 gene carriers and 20 controls will undergo 7T imaging
* blood and CSF sampling

We will compare change over time in preHD and control groups and model disease burden influence (an early natural history proxy) within the preHD group. These analyses will incorporate previous baseline measurements (providing three timepoints). We will create a data-driven natural history of pathological changes across the pre-clinical period in HD and estimate longitudinal models of age and CAG-dependence on the outcomes, providing a critical tool to increase power.

ELIGIBILITY:
Inclusion Criteria:

For the Healthy Control group, participants eligible are persons who meet the following criteria:

1. Are capable of providing informed consent and
2. Are capable of complying with study procedures and
3. Are aged between 18-47 years old and
4. Have no known family history of HD (gene negative); or
5. Have known family history of HD but have been tested for the huntingtin gene CAG expansion and are not at genetic risk for HD (CAG < 36*) (family control or community control)

For the Young Adult Premanifest HD group, participants eligible are persons who meet the following criteria:

1. Are capable of providing informed consent and
2. Are capable of complying with study procedures and
3. Are aged between 18-47 years old and
4. Have CAG expansion ≥ 40;
5. New participants must have a DBS <240

Exclusion Criteria:

Current use of investigational drugs or participation in a clinical drug trial within 30 days prior to study visit; or b. Current intoxication, drug or alcohol abuse or dependence; or c. If using any antidepressant, psychoactive, psychotropic or other medications or nutraceuticals used to treat HD, the use of inappropriate (e.g., non-therapeutically high) or unstable dose within 30 days prior to study visit; or d. Significant medical, neurological or psychiatric co-morbidity likely, in the judgment of the Principal Investigator, to impair participant's ability to complete essential study procedures; or e. Predictable non-compliance as assessed by the Principal Investigator; or f. Inability or unwillingness to undertake any of the essential study procedures; or g. Needle phobia: or h. Contraindication to MRI, including, but not limited to, MR-incompatible pacemakers, recent metallic implants, foreign body in the eye or other indications, as assessed by a standard pre-MRI questionnaire;or i. Pregnant (as confirmed by urine pregnancy test); or j. Claustrophobia, or any other condition that would make the subject incapable of undergoing an MRI.

For CSF collection:

1. Needle phobia, frequent headache, significant lower spinal deformity or major surgery; or
2. Antiplatelet or anticoagulant therapy within the 14 days prior to sampling visit, including but not limited to: aspirin, clopidogrel, dipyridamole, warfarin, dabigatran, rivaroxaban and apixaban; or
3. Clotting or bruising disorder; or
4. Screening blood test results outside the clinical laboratory's normal range for the following: white cell count, neutrophil count, lymphocyte count, haemoglobin (Hb), platelets, prothrombin time (PT) or activated partial thromboplastin time (APTT); or
5. Screening blood test results for C-reactive protein (CRP)>2× upper limit of normal; or
6. Exclusion during history or physical examination, final decision to be made by the Principal Investigator; including but not limited to:

i any reason to suspect abnormal bleeding tendency, e.g. easy bruising, petechial rash; or ii any reason to suspect new focal neurological lesion, e.g. new headache, optic disc swelling, asymmetric focal long tract signs; or iii any other reason that, in the clinical judgment of the operator or the Principal Investigator, it is felt that lumbar puncture is unsafe.

For Optional 7T MRI and MEG

1. Contraindication to MRI, including, but not limited to, MR-incompatible pacemakers, recent metallic implants, foreign body in the eye or other indications, as assessed by a standard pre-MRI questionnaire; or
2. Pregnant (as confirmed by urine pregnancy test); or
3. Claustrophobia, or any other condition that would make the subject incapable of undergoing an MRI; or
4. Tattoos that fall above the line defined by the crease of the elbow or on the genitals.

Ages: 18 Years to 47 Years | Sex: All
Age Groups: Adult
Study Population: Young adult Huntington's disease gene carriers and age-, sex- and education-matched controls between the ages of 18 and 47
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Brain volume in ml | Baseline, 4.5 years, 6 years
  Global and regional measures of brain volume
Biofluids in grams per litre | Baseline, 4.5 years, 6 years
  Blood and CSF measures
Cognition (raw scores) | Baseline, 4.5 years, 6 years
  Cognitive tests including CANTAB and EMOTICOM

CONTACTS AND LOCATIONS:
Locations (1):
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Scahill RI, Farag M, Murphy MJ, Hobbs NZ, Leocadi M, Langley C, Knights H, Ciosi M, Fayer K, Nakajima M, Thackeray O, Gobom J, Ronnholm J, Weiner S, Hassan YR, Ponraj NKP, Estevez-Fraga C, Parker CS, Malone IB, Hyare H, Long JD, Heslegrave A, Sampaio C, Zhang H, Robbins TW, Zetterberg H, Wild EJ, Rees G, Rowe JB, Sahakian BJ, Monckton DG, Langbehn DR, Tabrizi SJ. Somatic CAG repeat expansion in blood associates with biomarkers of neurodegeneration in Huntington's disease decades before clinical motor diagnosis. Nat Med. 2025 Mar;31(3):807-818. doi: 10.1038/s41591-024-03424-6. Epub 2025 Jan 17. PMID 39825149

DOCUMENTS (4):
  • Study Protocol (2023-09-07): https://cdn.clinicaltrials.gov/large-docs/19/NCT06391619/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT06391619/SAP_001.pdf
  • Informed Consent Form: Gene carrier (2023-09-07): https://cdn.clinicaltrials.gov/large-docs/19/NCT06391619/ICF_002.pdf
  • Informed Consent Form: Control (2023-09-07): https://cdn.clinicaltrials.gov/large-docs/19/NCT06391619/ICF_003.pdf